CLINICAL TRIAL: NCT04072874
Title: Evaluation of the Safety and Clinical Activity of Curaleish Lotion and Cream in the Topical Treatment of Cutaneous Leishmaniasis in Colombia
Brief Title: Evaluation of the Safety and Clinical Activity of Curaleish in the Topical Treatment of Cutaneous Leishmaniasis.
Acronym: Curaleish
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Tthe study is in the approval phase by local regulatory authorities
Sponsor: Universidad de Antioquia (Other)
Collaborators: INNOVATION CORPORATION FOR THE DEVELOPMENT OF PRODUCTS FOR TROPICAL DISEASES (CIDEPRO) (Unknown); Comprehensive Strategy for the Control of Leishmaniasis in Colombia (Unknown)
Responsible Party: Principal Investigator, Ivan Darío Vélez Bernal MD. MSc.. PhD., Full professor Faculty of Medicine - PECET, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEC02_2019
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2020-11

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Leishmaniasis; Curaleish
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

STUDY DESIGN:
Intervention Model Description: An Open-label, Randomized, Non-comparative, Two-arm Exploratory study. After all the screening evaluations have been completed, the principal investigator or his designee will confirm the patient's eligibility on Day 1, and the randomization will be determined by IWRS where randomized identification of the patient will be provided.
  The treatment allocation will be performed according to a computer-generated random code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Régimen 1 (Active Comparator): * Regimen 1: Curaleish lotion applied three times a day in combination with Curaleish cream applied two times a day for 4 weeks.
  * For both treatments, the patient applies Curaleish lotion in the morning, afternoon, and evening, that is to say, three times a day. And Curaleish cream in the morning and afternoon, that is, twice a day.
  Interventions: Drug: Experimental topical (Curaleish Topical)
- Régimen 2 (Active Comparator): * Regimen 2: Curaleish lotion applied three times a day in combination with Curaleish cream applied two times a day for 6 weeks.
  * For both treatments, the patient applies Curaleish lotion in the morning, afternoon, and evening, that is to say, three times a day. And Curaleish cream in the morning and afternoon, that is, twice a day.
  Interventions: Drug: Experimental topical (Curaleish Topical)

INTERVENTIONS:
Drug: Experimental topical (Curaleish Topical) — Curaleish is a formulation in lotion and cream. Curaleish lotion and Curaleish cream will be applied topically by each participant in all lesion until day 28 or 42, depending on the regimen to be evaluated. Study staff will be closely observing the safety assessment. The application until Day 28 or 42 will continue, even if the lesion has shown 100% re-epithelization before day 28 or day 42.
  Other Names: Curaleish Topical

SUMMARY:
Cutaneous Leishmaniasis (CL) is a parasitic disease caused by more than 15 different species of the protozoan parasite Leishmania. The CL usually begins with a papule at the site of the sandfly bite, increasing in size to form a nodule that ulcerates in a period of 1 to 3 months.

The exact incidence of CL is not known. An estimated 1.2 million cases/year in approximately 102 countries worldwide suffer from different forms of CL. Among the different parasites that cause CL, L.tropica in the Old World and L.braziliensis in the New World are considered to be the most important due to the difficulty of healing, the public importance and the severity of the disease.

Pentavalent antimony remains the first choice drug for the treatment of CL and the evidence to support its use is sometimes based on qualitative, retrospective and uncontrolled observations, with only some controlled clinical studies. Antimonials are widely used despite their toxicity, difficulty in the route of administration, and high cost.

Miltefosine (hexadecylphosphocholine), an oral medication that has proven effective for some types of Leishmania, is potentially teratogenic, is contraindicated during pregnancy and requires appropriate counseling for female patients of childbearing age.

DETAILED DESCRIPTION:
Curaleish is a topical formulation in lotion and cream that contains natural extracts (hydroalcoholic and glycolic for lotion and cream, respectively) of the branches (stems and leaves) of the Caesalpinia spinosa tree known as "Tara" or "Davidivi" , which was developed by Bionest SAS, Duitama, Colombia.

The product is currently manufactured by Biohealthy SD S.A.S in accordance with Colombian Good Manufacturing Practices (BPM) and evaluated by PECET following the international standardized animal protocols and models of OECD.

The development of a topical formulation of Curaleish is intended to offer a treatment to be applied locally in the lesion of the LC, with a high antiparasitic effect. The formulation of Curaleish lotion and Curaleish cream containing natural extracts, started from the activity demonstrated in In vitro for the hydroalcoholic extract of C. espinosa (EC50 = 18.4 ± 1.3 µg / mL) and a low cytotoxicity evidenced by an LC50 of 135.6 ± 0.7, 183.3 ± 1.1 and 136.6 ± 7.4 µg / mL in human liver cells HepG2, human macrophages U937 and peritoneal hamster macrophages, respectively, and a selectivity index of 9.41, 9.96 and 7.42, respectively. This activity was validated in in vivo studies in hamsters experimentally infected with L. braziliensis. Applying the cream alone twice a day for 28 days produced a cure in 83% and fails in 17%. On the other hand, the lotion applied once a day for 28 days showed cure in 67% and relapse in 33%. When the lotion was used in combination twice a day and the cream once a day for 28 days, 100% cure was achieved, which occurred early in most hamsters, this is at the end of the treatment.

Accelerated stability tests for 3 months and natural stability (6 months) under Zone IV conditions of the ICH (conditions 25ºC / 60% RH, 30ºC / 65% RH, 30ºC / 75% RH and 40ºC / 75% RH) have shown that the product meets the criteria required for physical and microbiological analysis, established by the United States Pharmacopeia (USP). These parameters are for the cream: density 0.957 ± 0.000 g / mL for the cream and 0.958 ± 0.000 g / mL for the lotion; Extensibility area 123.24 ± 19.64 mm2 for the cream; pH of 6.69 ± 0.115 for the cream and 4.82 ± 0.017 for the lotion; <104 CFU of total aerobes and <103 CFU / mL for molds and yeasts.

Weight, clinical appearance and behavior data, as well as histological studies obtained from preclinical acute dermal toxicity tests as well as cellular viability data obtained in skin irritation / corrosion tests for Curaleish lotion and cream, executed according With the OECD guidelines, it was concluded that skin contact with Curaleish products does not generate toxic effects at the local level (application site) or at the systemic level, so it can be considered as safe for use.

An exploratory study to assess the safety, and to determine whether the Curaleish topical cream when the lotion is applied three times a day in combination with the cream, applied twice a day for 4 weeks showed that it is 83% effective for treatment of Colombian subjects with uncomplicated LC. 25 of 30 patients managed to cure between 1.5 and 3 months after the end of Curaleish treatment.

The development of a topical formulation of Curaleish is intended to offer a treatment to be applied locally in the lesion of the CL, with a high antiparasitic effect. Skin irritation/corrosion tests for Curaleish lotion and cream, performed following the guidelines of the OECD, allowed to conclude that skin contact with Curaleish products does not generate toxic effects locally, or at a systemic level, therefore they can be considered safe for use.

Main Objectives To assess the safety and tolerability of two Curaleish regimens administered topically in individuals with uncomplicated CL.

The two regimes to evaluate are:

* Regimen 1: Curaleish lotion applied three times a day in combination with Curaleish cream applied two times a day for 4 weeks.
* Regimen 2: Curaleish lotion applied three times a day in combination with Curaleish cream applied two times a day for 6 weeks.

Secondary Objectives Evaluate the safety of Curaleish (frequency and severity of adverse events (AEs)). Other secondary efficacy objectives include the assessment of the condition of the lesions over time up to 100% re-epithelialization of the ulcerated lesions and the proportion of individuals with 100% re-epithelization of not ulcerated lesions over time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 - 60 years.
* Patient with confirmed parasitological diagnosis of CL in at least one lesion, performed at least through the following methods: 1) microscopic identification of amastigotes in tissue of the lesion; 2) Leishmania diagnose through PCR; 3) positive culture for promastigotes.
* Patient with a lesion that meets the following criteria:

  . Ulcer or nodule with a maximum size of 4 cm (the largest diameter).
* Not located in the ear, face, near mucous membranes, joints, or in places that, in the opinion of the PI, the study medication is difficult to apply topically.
* Patient with a maximum of four CL lesions.
* The duration of the lesion is less than three months according to the patient's history.
* The patient is able to give written informed consent.
* Patients whom the investigator believes are able to understand and are willing to comply with the requirements of the protocol.

Exclusion Criteria:

Patients who meet some of the following criteria must be excluded from the study:

* Women with positive pregnancy test during the screening process, or who are lactating; or women of childbearing age who do not agree to take contraceptives during treatment and until Day 45.
* The subject has a history of significant medical conditions or treatments that may interact negatively or positively with the topical treatment of Leishmaniasis, including any immune compromise condition.
* Within eight weeks (56 days) of beginning the study treatments, having received treatment for Leishmaniasis through any medication, including Glucantime that probably, in the opinion of the principal investigator (PI), might modify the course of the infection by Leishmania.
* Based on physical examinations performed, they have been diagnosed, or a diagnosis of Mucocutaneous Leishmaniasis is suspected.
* Known history or suspected hypersensitivity or idiosyncratic reactions to the study medication.
* Patients who do not wish to attend study appointments or who cannot keep up with follow-up visits for up to 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
post treatment (healing) | day 180
  Healing: initial healing * without relapse and/or mucous commitment for the post-treatment evaluation of Day 180.
  *Initial healing: defined as 100% re-epithelialization of the lesion(s) following Day 90 post-treatment.

SECONDARY OUTCOMES:
2. Days 28 and 42, respectively, depending on the duration of each treatment group. (Adverse events) | 28 days and 42 days
  Adverse events (AEs) will be evaluated according to the seriousness, temporal relationship, relationship with the study medication, and severity. The recording will be carried out through clinical examination, telephone calls, and through the completion of the subject's diary.
  The local AEs that will be evaluated are:
  1. Erythema
  2. Burning
  3. Pain
  4. Pruritus
  5. Irritation
  The following evaluations will be made:
  * Frequency and severity (Mild, Moderate, Severe) of AEs by treatment group.
  * Status (area of lesions, induration, erythema, etc.) in each measurement. Additionally, before starting treatment and at the end of it, renal (creatinine) and liver function (transaminases) tests will be performed on volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan D Velez, Principal Investigator — Director PECET
Locations (1):
- Program for Research and Control in Tropical Diseases - PECET, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blum J, Lockwood DN, Visser L, Harms G, Bailey MS, Caumes E, Clerinx J, van Thiel PP, Morizot G, Hatz C, Buffet P. Local or systemic treatment for New World cutaneous leishmaniasis? Re-evaluating the evidence for the risk of mucosal leishmaniasis. Int Health. 2012 Sep;4(3):153-63. doi: 10.1016/j.inhe.2012.06.004. PMID 24029394
- [Background] Blum J, Desjeux P, Schwartz E, Beck B, Hatz C. Treatment of cutaneous leishmaniasis among travellers. J Antimicrob Chemother. 2004 Feb;53(2):158-66. doi: 10.1093/jac/dkh058. Epub 2004 Jan 16. PMID 14729756
- [Background] Soto J, Rea J, Balderrama M, Toledo J, Soto P, Valda L, Berman JD. Efficacy of miltefosine for Bolivian cutaneous leishmaniasis. Am J Trop Med Hyg. 2008 Feb;78(2):210-1. PMID 18256415
- [Background] WHO technical report series; no. 949. Control of the leishmaniasis: report of a meeting of the WHO Expert Committee on the Control of Leishmaniases, Geneva, 22-26 March 2010.
- [Background] Silva NS, Muniz VD. [Epidemiology of American tegumentary leishmaniasis in the State of Acre, Brazilian Amazon]. Cad Saude Publica. 2009 Jun;25(6):1325-36. doi: 10.1590/s0102-311x2009000600015. Portuguese. PMID 19503963
- [Background] Almeida OL, Santos JB. Advances in the treatment of cutaneous leishmaniasis in the new world in the last ten years: a systematic literature review. An Bras Dermatol. 2011 May-Jun;86(3):497-506. doi: 10.1590/s0365-05962011000300012. English, Portuguese. PMID 21738967
- [Background] Tiuman TS, Santos AO, Ueda-Nakamura T, Filho BP, Nakamura CV. Recent advances in leishmaniasis treatment. Int J Infect Dis. 2011 Aug;15(8):e525-32. doi: 10.1016/j.ijid.2011.03.021. Epub 2011 May 24. PMID 21605997
- [Background] Herwaldt BL. Leishmaniasis. Lancet. 1999 Oct 2;354(9185):1191-9. doi: 10.1016/S0140-6736(98)10178-2. PMID 10513726
- [Background] Velez I, Lopez L, Sanchez X, Mestra L, Rojas C, Rodriguez E. Efficacy of miltefosine for the treatment of American cutaneous leishmaniasis. Am J Trop Med Hyg. 2010 Aug;83(2):351-6. doi: 10.4269/ajtmh.2010.10-0060. PMID 20682881
- [Background] Croft SL, Seifert K, Yardley V. Current scenario of drug development for leishmaniasis. Indian J Med Res. 2006 Mar;123(3):399-410. PMID 16778319
- [Background] Pearson, R. D., and A. de Querez Sousa. 1995 Leishmania species: visceral (kala-azar), cutaneous, and mucosal leishmaniaisis. p. 2428-2442. In G. L. Mandell, J. E. Bennett, and R. Dolin (ed.) Principles and practice of infectious diseases. Churchill Livingstone, New York, N.Y.
- [Background] Votypka J, Kasap OE, Volf P, Kodym P, Alten B. Risk factors for cutaneous leishmaniasis in Cukurova region, Turkey. Trans R Soc Trop Med Hyg. 2012 Mar;106(3):186-90. doi: 10.1016/j.trstmh.2011.12.004. Epub 2012 Jan 26. PMID 22284721
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Reveiz L, Maia-Elkhoury AN, Nicholls RS, Romero GA, Yadon ZE. Interventions for American cutaneous and mucocutaneous leishmaniasis: a systematic review update. PLoS One. 2013 Apr 29;8(4):e61843. doi: 10.1371/journal.pone.0061843. Print 2013. PMID 23637917
- [Background] Lee SA, Hasbun R. Therapy of cutaneous leishmaniasis. Int J Infect Dis. 2003 Jun;7(2):86-93. doi: 10.1016/s1201-9712(03)90002-6. PMID 12839708
- [Background] Lopez L, Robayo M, Vargas M, Velez ID. Thermotherapy. An alternative for the treatment of American cutaneous leishmaniasis. Trials. 2012 May 17;13:58. doi: 10.1186/1745-6215-13-58. PMID 22594858
- [Background] Organizacion Panamerica de la Salud, OPS. Leishmaniasis en las Americas: Recomendaciones para el tratamiento. 2013. http://www.paho.org/hq/index.php?option=com_docman&task=doc_view&gid=22226&Itemid
- [Background] Velasco-Castrejon O, Walton BC, Rivas-Sanchez B, Garcia MF, Lazaro GJ, Hobart O, Roldan S, Floriani-Verdugo J, Munguia-Saldana A, Berzaluce R. Treatment of cutaneous leishmaniasis with localized current field (radio frequency) in Tabasco, Mexico. Am J Trop Med Hyg. 1997 Sep;57(3):309-12. doi: 10.4269/ajtmh.1997.57.309. PMID 9311641